CLINICAL TRIAL: NCT04909294
Title: Multicenter Phase II Study Evaluating the Efficacy and Safety of a Stereotaxic Prostatic Radiotherapy Delivered on Linac MRI, With Integrated Boost in the Case of an Index Tumor, in Patients With Prostate Adenocarcinoma of Favorable, Intermediate or Risky Risk. High Risk Very Localized.
Brief Title: Evaluation of the Efficacy and the Safety of a Stereotaxic Prostatic Radiotherapy Delivered With Linac MRI, in Patients With Prostate Adenocarcinoma
Acronym: STEREO-RML
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STEREO-RML
Record Dates: First submitted 2021-05-21; First posted 2021-06-01 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Adenocarcinoma of the Prostate
Keywords: radiotherapy
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- stereotaxic external radiation therapy (Experimental)
  Interventions: Radiation: Stereotactic Radiotherapy with Linac MRI

INTERVENTIONS:
Radiation: Stereotactic Radiotherapy with Linac MRI — 38 Gy in 4 fractions of 9.5 Gy over the entire prostate,
  +/- 2 Gy in 4 fractions of 0.5 Gy as an integrated boost on the index tumor if it is visible on diagnostic multiparametric MRI (PIRADS-V2 score 4 or 5) and on planning MRI performed on Linac MRI.

SUMMARY:
Stereotaxic prostatic radiotherapy on Linac MRI, with monitoring of movements of the pelvic organs per fraction on the prostate in real time, in 4 sessions, with integrated boost on the index tumor (if it is visible on the diagnostic MRI), could reduce the digestive, urinary and sexual toxicities accumulated at 5 years and guarantee excellent local tumor control, for patients with localized prostate cancer, with a favorable prognosis, intermediate or very local high risk, according to the D'Amico classification.

The benefits that patients participating in this research could obtain are:

* Better disease control efficiency
* A reduction in the duration of treatment to 4 radiotherapy sessions (2 weeks maximum) instead of 40 sessions (8 weeks) for usual treatment.
* Avoid the risks associated with the implantation of prostate markers necessary for stereotaxic radiotherapy on a standard accelerator (anesthetic risks, infectious risks, hemorrhagic risks, pain risks)
* Better quality of life

ELIGIBILITY:
Inclusion Criteria:

1. prostate adenocarcinoma
2. WHO performance index ≤ 1
3. Patient presenting one of the following cases:

   * Low risk: ≤ T2a and Gleason 6 (3 + 3) and PSA <10 ng / ml
   * Intermediate risk: T2b-T2c or Gleason 7 or PSA <15 ng / ml
   * High localized risk: T3a and Gleason ≤7 and PSA <15 ng / ml
4. Disease presenting a risk of lymph node involvement <15%
5. Absence of pelvic or lumbar aortic lymphadenopathy
6. Absence of bone or visceral metastasis
7. IPSS score <15 or ≤ 7
8. Prostate volume estimated by MRI or ultrasound < 90cc
9. If hormonotherapy, hormone therapy must not have started for more than 60 days before inclusion.
10. Absence of prior pelvic radiotherapy
11. No surgical treatment for prostate cancer

Exclusion Criteria:

1. Prostate cancer of histology other than adenocarcinoma
2. Contraindication to MRI including, but not limited to, patients with a pacemaker or defibrillator
3. Patient diagnosed N1 during imaging workup or pN1
4. Serum PSA level ≥ 15 ng / ml
5. IPSS score ≥ 15 or IPSS score> 7 if alpha blocking urological treatment in progress
6. Prostate volume estimated on MRI or ultrasound> 90 cc
7. Involvement of seminal vesicles on MRI
8. History of cancer in the 5 years preceding entry into the trial
9. History of transurethral resection of the prostate less than 6 months compared to the expected date of start of radiotherapy
10. rectal surgery
11. pelvic irradiation
12. Patient treated with antineoplastic or medication which may include Methotrexate
13. Hormone therapy started for more than 60 days at the time of inclusion
14. Severe uncontrolled hypertension
15. Patient followed or treated for severe or unstable angina, or having presented a myocardial infarction in the 6 months preceding the randomization
16. Patient on immunosuppressant
17. Patient with known hypersensitivity to gadoteric acid, meglumine or any drug containing gadolinium

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Late gastrointestinal and urinary toxicity grade ≥ 2 | 5 years
  toxicities graded according to the NCI-CTCAE-V5.0

CONTACTS AND LOCATIONS:
Overall Officials: Magali QUIVRIN, Principal Investigator — Centre Georges François Leclerc
Locations (1):
- Centre Georges François Leclerc, Dijon, France